CLINICAL TRIAL: NCT04413500
Title: iMedA: Improving MEDication Adherence Through Person Centered Care and Adaptive Interventions
Brief Title: iMedA: Improving MEDication Adherence Through Person-Centered Care and Adaptive Interventions
Acronym: iMedA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Halmstad University (Other)
Collaborators: Region Halland (Other)
Responsible Party: Principal Investigator, Kobra Etminani, Assistant Professor at CAISR, department of ISDD, School of ITE, HH, Halmstad University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-04617
Record Dates: First submitted 2020-05-22; First posted 2020-06-04 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Hypertension
Keywords: hypertension; digital intervention; adaptive intervention
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adaptive intervention (Experimental): The patients will receive various adaptive digital interventions through mobile app.
  Interventions: Behavioral: Reminder; Behavioral: Educational message; Behavioral: Motivational messages; Behavioral: showing trends

INTERVENTIONS:
Behavioral: Reminder — A reminder to take the anti-hypertension medication with adjustable frequency.
Behavioral: Educational message — An educational message to increase the knowledge about various facts around hypertension. The short messages are supposed to be sent based on the patient's needs.
Behavioral: Motivational messages — The motivational short messages to increase the motivational levels.
Behavioral: showing trends — Short messages contain different trends of medication intake rate, BP, physical activity rate, and so on.

SUMMARY:
The aim of this study is to design, implement, and evaluate an adaptive personalized digital intervention, to be delivered through a mobile application, to increase medication adherence and self-care management for persons with hypertension. This is a collaborative project between Halmstad University and Region Halland in Halland county, Sweden.

The project is divided into three steps: 1)Focus groups 2)pilot study 3)Longitudinal study. The design of the study is influenced by the Intervention Mapping technique, which is used for the design and development of health promotion programs. The investigators first conducted a systematic review in order to detect the determinants, behaviors to change, and implemented digital strategies in the previous studies. The result was drawn in the Matrix of Change Objectives to facilitate the mapping. Then through focus groups, the investigators are going to ascertain the needs of the Swedish context. Through what has been learned with these findings, digital interventions will be designed and developed to be delivered via mobile application. A pilot study is considered then to evaluate the feasibility and usability testing of digital intervention. Finally, a longitudinal study is designed to evaluate the effectiveness of the digital intervention in the longer term. The design is proposed to be an interrupted time series (ITS) approach which is considered to be the strongest quasi-experimental design that can be used to evaluate the effectiveness of an intervention.

DETAILED DESCRIPTION:
The design of the digital intervention module is considered to follow the just-in-time adaptive intervention framework (JITAI). JITAI is an intervention design aiming to provide the right type/amount of support, at the right time, by adapting to an individual's circumstances. It has enormous potential for promoting health behavior change, which in this study is supposed to be medication compliance. Based on the JITAI's conceptual model, there are the following components:

1. Decision points (DP) DP is a time when an intervention decision is made. Considering the nature of JITAIs which are delivered through mobiles, DPs are much more rapidly than is standard interventions. In iMedA, DP is considered to be daily and accompanied by the time of medication intake question, i.e. "Did the participant take the anti-hypertensive medication today?".
2. Intervention options (IO) IOs are a set of possible interventions that are going to be delivered at DPs. In JITAI, IOs can be various types of support (information, advice, feedback, etc), source of support (mobile, nurse, physician, etc), amounts of support (intensity, dose, etc), type of media/channel (phone call, SMS, etc).

   From the conducted literature review, the investigators summarised all types of digital interventions to hypertensive patients as:
   * Reminders for medication intake (daily), BP measurement (monthly), PA (biweekly)
   * Informational contents regarding hypertension and all its facts, consequences, treatments, risks, medications and side-effects, lifestyle, and so on (text, videos, etc)
   * Trends on medication intake/PA/BP/etc
   * Motivational messages
3. Distal outcomes (DO) DO is the ultimate goal that the intervention is trying to achieve. In iMedA, the investigators considered primary and secondary DOs. Primarily the investigators aim at improving medication adherence. Then in the long term, blood pressure control is considered as secondary DOs besides the increased quality of life, assessment of the lifestyle behavior (smoking, alcohol consumption, physical activity, and food intake), and communicative and critical health literacy.

   In order to measure MA, the investigators consider (1) self-reported medication intake through a mobile app; (2) MUAH-16 which is a medication adherence questionnaire for hypertension; and (3) pickups from pharmacies. The self-reported values are supposed to be collected every day. MUAH-16 is measured pre- and post- intervention.

   BP is considered to be measured every month. There are automatic devices in every primary care center that people can go and measure their BP free of charge.

   QoL and HL are measured through EQ5D and HL respectively and pre- and post- intervention. Lifestyle assessments are measured (bi)weekly through self-report values.
4. Proximal outcomes (PO) POs are the short-term goals of the interventions. They can be mediators and/or intermediate measures of the DOs. Medication intake rate is considered to be the main PO, which is measured daily. Physical activity rate which is measured (bi)weekly is another PO.

   Since most of the contents are educational and they try to increase the hypertension knowledge of the participants, the investigators will add a PO to measure how much their knowledge has increased. The investigators consider two methods to measure it. First, after showing the content, the investigators will ask "Did the participant know …?". Second, a simple gamification test will be designed to be delivered biweekly.

   To prevent poor adherence to the interventions, it is recommended to define a few POs related to intervention engagement and fatigue. Therefore, the investigators consider the number of clicked interventions, number of watched videos, like/dislike feedbacks per each intervention as POs related to intervention adherence and retention.
5. Tailoring variables (TV) TVs are information about the participant that are used to decide when to provide which intervention. In other words, they are used to personalise the interventions and make them adaptive to the individual's circumstances. They can be measured actively or passively or both. Active assessments require an individual's engagement in measuring, for example through self-reports, while passive assessments require minimal/no individual engagement, for example through mobile phone's sensors. POs are often used as TVs.

   From baseline information, a few TVs can be selected including alcohol consumption, smoking, specific diet (vegetarian, vegan, etc), age, and gender, in order to personalise the interventions.

   All of the POs are also considered as TVs. From the MUAH-16 questionnaire, the investigators start to know more about individual's beliefs, barriers and behaviour about medication adherence. It has four subscales regarding (1)positive attitude towards healthcare and medication; (2) lack of discipline; (3) aversion towards medication; and (4) active coping with health problems. Each subscale contains four questions. At the beginning of the intervention, MUAH-16 questions are used as TVs. Then during the intervention period, and based on the previously delivered informational contents to the individual, the answers to "Did the participant know …?" questions will be used as TVs.
6. Decision rules (DR) DRs are the adaptation engine of JITAIs. They are used to determine which IO to deliver to whom and when. They are the links between IOs and TVs.

DRs in iMedA will be probabilistic rules from experts modified by "suggestions" from reinforcement learning.

ELIGIBILITY:
Inclusion Criteria:

* aged 40-70 years old
* have hypertension diagnosis (i.e. ICD 10 codes from I10 to I16 in the person's medical history) for 1 year or more and have prescribed medications;
* not receiving medication with unit-dose packaged (Apodos);
* no previous stroke or myocardial infarction;
* no psychological disorder or cognitive impairment;
* no pregnancy-induced hypertension;
* no insulin treatment;
* no kidney disease defined as glomerular filtration rate (GFR) <60 ml/min

Exclusion Criteria:

* have no own smartphone
* not understanding the Swedish language both spoken and written

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
change from baseline medication adherence score at 6 months | 6 months
  medication adherence score (MA) measured through the Maastricht Utrecht Adherence in Hypertension (MUAH-16) questionnaire.
  The higher score is correlated to better medication adherence. MUAH-16 has 4 subscales: 2 of them measures positive and the other 2 measures negative aspects of medication adherence. Therefore, we consider a positive score for the 2 positive subscales and negative scores to the negative ones. The result will be the final score showing the medication adherence score of the participant.
  The answers are supposed to be on a 7-point Likert scale (1: completely disagree and 7:completely agree). Therefore, the max score will be 48 and the min score will be -48.
  Based on the previous study, there has been shown a correlation between having a higher score and higher medication adherence.

SECONDARY OUTCOMES:
change from baseline Blood pressure at 6 months | 6 months
  Systolic and diastolic Blood Pressure (BP). The lower BP the better outcome.
change from baseline health literacy score at 6 months | 6 months
  health literacy (HL) measured through the Communicative and Critical Health Literacy Scale.
  We expect to see an increase in HL through time, therefore the higher HL the better outcome.
  Considering the 5-point Likert scale , the max score will be 25 and the min score will be 5.
change from baseline Quality of Life at 6 months | 6 months
  quality of life measured through the EuroQol- 5 Dimension (EQ5D) instrument. The higher score the better outcome.
  The answers to each of the five dimensions is between 1-3 scale. The EQ-VAS scale is between 0-100.

OTHER OUTCOMES:
medication intake rate | through study completion, an average of 6 months
  self-reported medication intake. We expect to see an increase in the medication intake rate.
physical activity | through study completion, an average of 6 months
  physical activity rate. We expect to observe a higher physical activity rate.
change from baseline medication pickups from pharmacies at 6 months | 6 months
  check the anti-hypertensive medication pickups from pharmacies. We expect that the pickups from pharmacies will increase.

CONTACTS AND LOCATIONS:
Overall Officials: Kobra Etminani, Principal Investigator — Halmstad University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nahum-Shani I, Smith SN, Spring BJ, Collins LM, Witkiewitz K, Tewari A, Murphy SA. Just-in-Time Adaptive Interventions (JITAIs) in Mobile Health: Key Components and Design Principles for Ongoing Health Behavior Support. Ann Behav Med. 2018 May 18;52(6):446-462. doi: 10.1007/s12160-016-9830-8. PMID 27663578
- [Background] Cabral AC, Castel-Branco M, Caramona M, Fernandez-Llimos F, Figueiredo IV. Developing an adherence in hypertension questionnaire short version: MUAH-16. J Clin Hypertens (Greenwich). 2018 Jan;20(1):118-124. doi: 10.1111/jch.13137. Epub 2017 Nov 24. PMID 29171719
- [Background] Wagner AK, Soumerai SB, Zhang F, Ross-Degnan D. Segmented regression analysis of interrupted time series studies in medication use research. J Clin Pharm Ther. 2002 Aug;27(4):299-309. doi: 10.1046/j.1365-2710.2002.00430.x. PMID 12174032
- [Result] Etminani K, Tao Engstrom A, Goransson C, Sant'Anna A, Nowaczyk S. How Behavior Change Strategies are Used to Design Digital Interventions to Improve Medication Adherence and Blood Pressure Among Patients With Hypertension: Systematic Review. J Med Internet Res. 2020 Apr 9;22(4):e17201. doi: 10.2196/17201. PMID 32271148
- [Derived] Etminani K, Goransson C, Galozy A, Norell Pejner M, Nowaczyk S. Improving Medication Adherence Through Adaptive Digital Interventions (iMedA) in Patients With Hypertension: Protocol for an Interrupted Time Series Study. JMIR Res Protoc. 2021 May 12;10(5):e24494. doi: 10.2196/24494. PMID 33978593